CLINICAL TRIAL: NCT02084472
Title: Accessible and Affordable Moisturizers for Atopic Eczema: the 2am Atopic Eczema Study
Brief Title: Accessible and Affordable Moisturizers for Atopic Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Red Cross War Memorial Childrens Hospital (Other)
Responsible Party: Principal Investigator, Dr Carol Hlela, Dermatologist, Red Cross War Memorial Childrens Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 146/2013
Record Dates: First submitted 2014-03-03; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Childhood Atopic Dermatitis
Keywords: atopic eczema; moisturisers; alternatives; affordable
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study 1: aqueous cream and baby oil (Active Comparator): enrolled patients in this arm use either aqueous cream or baby oil as a soap substitute
  Interventions: Other: Baby oil
- study 2: emulsifying ointment and cetomacrogol (Active Comparator): patients in this study arm continue to use emulsifying ointment and cetomacrogol as a moisturiser, the current standard of care in our institution
  Interventions: Other: petroleum jelly; Other: Glycerine:petroleum jelly 2:1

INTERVENTIONS:
Other: Baby oil — patient in study 1, arm B washed unscented liquid paraffin (baby oil) in place of aqueous cream
  Other Names: unscented liquid paraffin
  Arms: study 1: aqueous cream and baby oil
Other: petroleum jelly — patients in this arm, use petroleum jelly (vaseline), replacing emulsifying ointment as a moisturiser
  Arms: study 2: emulsifying ointment and cetomacrogol
Other: Glycerine:petroleum jelly 2:1 — patients in this arm use glycerine and petroleum jelly mixed at a ratio of 2:1 in place of cetomacrogol as a moisturiser
  Arms: study 2: emulsifying ointment and cetomacrogol

SUMMARY:
Aqueous (EUA) cream, cetomacrogol (CMG) and emulsifying ointment (HEB) are in South Africa's essential drug list (EDL) but are not available to most rural patients. To assess whether accessible moisturizers can be used as alternatives in atopic eczema (AD), a randomized controlled trial of patients with mild-to-moderate AD, aged 1-12 years was conducted. Two separate sub-studies were conducted using a randomized controlled single (assessor) blind trial design. Study 1 compared UEA vs. liquid paraffin (unscented baby oil) for baths, all patients used HEB as moisturiser. In Study 2, 4 moisturisers were compared -HEB, CMG, petroleum jelly and petroleum jelly/Glycerine (2:1). Assessments (SCORAD, POEM, NESS and IQDOL) carried out at baseline, week 4, 8 and 12. Routine topical steroids and antihistamines were continued as prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Atopic dermatitis as defined by the united kingdom (UK) Working party Diagnostic Criteria
* Atopic Dermatitis patient with mild to moderate stable atopic eczema with parents/guardians willing and able to apply study moisturizers as directed and commit to attend all visits.

Exclusion Criteria:

* Less than 1 year of age
* Patients with atopic dermatitis treated with systemic preparations

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in the validated SCORing Atopic Dermatitis(SCORAD) | Baseline, week 4, 8 and week 12
  Change in the validated SCORing Atopic Dermatitis(SCORAD) and two other validated clinical scores (Nottingham Atopic Eczema Severity Score(NESS) and Patient Oriented Eczema Measure(POEM) were used to measure the extent/severity of AD. A validated quality-of-life form using the infants dermatitis quality of life (IDQOL) scale was completed by each care-giver at each visit.

SECONDARY OUTCOMES:
Change in the patient quality-of-life as measured by the infants dermatitis quality of life (IDQOL) index at each visit. | Baseline, week 4, 8,12

CONTACTS AND LOCATIONS:
Overall Officials: Nonhlanhla Khumalo, MD, PhD, Study Director — University of Cape Town; Carol Hlela, MD, PhD, Principal Investigator — Red Cross War Memorial Children's Hospital
Locations (1):
- Red Cross War Memorial Children's Hospital, Cape Town, Western Cape, South Africa